CLINICAL TRIAL: NCT05043350
Title: Potential Therapeutic Outcome of Combined Antihistaminics Therapy in COVID 19 Patients
Brief Title: Combined Antihistaminics Therapy in COVID 19 Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Nasr City Insurance Hospital (Other Government)
Responsible Party: Principal Investigator, Samar Saad elDeen Azab, Professor of Pharmacology & Toxicology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACUCFPASURHDIRB2020110301REC43
Record Dates: First submitted 2021-09-11; First posted 2021-09-14 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Loratadine; Famotidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional group (Experimental): 107 patients will receive standard pharmacotherapy according to the treatment protocols of the National Committee of COVID-19 in addition to IV famotidine 40 mg twice daily (Manufactured by AMOUN Pharmaceutical Company) until the day of discharge + LORATIDINE (Manufactured by AMOUN Pharmaceutical Company)Oral: 10 mg once daily.
  Interventions: Drug: Loratadine; Drug: Famotidine
- Control group (Active Comparator): 107 patients will receive standard drug therapy according to the treatment protocols of the National Committee of COVID-19 in addition to IV famotidine 40 mg twice daily (Manufactured by AMOUN Pharmaceutical Company)
  Interventions: Drug: Famotidine

INTERVENTIONS:
Drug: Loratadine — 107 patients will receive standard pharmacotherapy according to the treatment protocols of the National Committee of COVID-19 in addition to IV famotidine 40 mg twice daily (Manufactured by AMOUN Pharmaceutical Company) until the day of discharge + LORATIDINE (Manufactured by AMOUN Pharmaceutical Company)Oral: 10 mg once daily.
  Arms: Interventional group
Drug: Famotidine — 107 patients will receive standard pharmacotherapy according to the treatment protocols of the National Committee of COVID-19 in addition to IV famotidine 40 mg twice daily (Manufactured by AMOUN Pharmaceutical Company) until the day of discharge + LORATIDINE (Manufactured by AMOUN Pharmaceutical Company)Oral: 10 mg once daily.

SUMMARY:
The use of antihistaminic medications could result in a significant immune modulation which may help in the treatment of cytokine storm of COVID-19.Thus, the aim of this study is to evaluate efficacy and safety of famotidine and loratadine combination in covid 19 treatment protocol.

DETAILED DESCRIPTION:
On admission to hospital, the patient will be diagnosed for suspected COVID-19 based primarily upon pulmonary symptoms, and will be confirmed positive for COVID-19 by RT-PCR diagnostic test and then will be located within a COVID-19 ward. According to Ministry of Health guidelines, moderate cases of COVID 19 will be identified if the Patient has pneumonia manifestations on radiology associated with symptoms (fever, cough, general weakness /fatigue, headache, sore throat, anorexia, diarrhea and vomiting) and / or leucopenia or lymphopenia.

Treatment will be initiated in ER with standard of care per admitting provider. Standard of care includes radiologic assessments, supplemental oxygen when necessary, and intravenous (IV) hydration when necessary. In addition to concomitant treatments like the antimalarial drug hydroxychloroquine, the anti-inflammatory drug dexamethasone (IV).plus, Famotidine 40 mg po twice daily and loratadine 10 mg po once daily (Interventional group) and Control group will receive standard drug therapy according to the treatment protocols of the National Committee of COVID-19 + Famotidine 40 mg twice daily po. The COVID-19 standard of care as provided by the ministry of health is attached in appendix1.Blood samples will be withdrawn from the patients at baseline and every 7 days to assess the following parameters using routine laboratory methods Complete blood picture: Lymphopenia, eosinopenia, neutrophil/lymphocyte ratio and platelet count, C-reactive protein and ferritin, lactate dehydrogenase (LDH), d-dimer Cardiac markers, IL-6, Procalcitonin, Prothrombin time, Activated partial thromboplastin time, Creatine kinase (CK), Glutamic-pyruvic transaminase (SGPT) and Urea, and serum creatinine to determine the incidence of organ failure Sample handling: Syringes used in sample withdrawal will be discarded in appropriate safety box and serum samples will be discarded in biohazards box. These biohazard waste will be sent to incinerators through the hospital laboratory as per hospital protocol.

Precaution against infections:

The principal investigator and all healthcare professional must wear full protective personal equipment (PPE) as per hospital protocol including full gown, full facial mask and safety gloves when in direct contact with patients for follow ups. These PPE are removed before the exit of COVID-19 ward and discarded as hazard waste. Disinfectant will be used by all personal before leaving the ward

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (>18 years old).
2. Confirmed COVId-19 infection with PCR.
3. Moderate covid patients who with Sp02 <92 %
4. CT chest infiltration more than 50 %
5. Presented to the hospital within 24 to 48 hours
6. CBC (WBCs may be normal or high or low with lymphocytopenia is present, decreased hemoglobin, neutrophilia with neutrophil/lymphocyte ratio > 3.1)

Exclusion Criteria:

1. Hepatic or renal failure: (Alanine transaminase or Aspartate transaminase >3 times above the normal limit)
2. History or evidence of long QT segment on Electrocardiogram,
3. Pregnancy or breast-feeding mother
4. Patient on mechanical ventilator.
5. Patient who received vaccine.
6. Patients receiving antidepressants, opioids, (e.g., anticonvulsants, clonazepam).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Assessment of number of patients who will need Mechanical ventillation | during hospital stay (Up to 28 days)
Assessment of the number of patients who will need vasopressor due to progression to shock | during hospital stay (Up to 28 days)

SECONDARY OUTCOMES:
Assessment of Duration (number of days) the patients will need oxygen support therapy | during hospital stay (Up to 28 days)
  the duration of oxygen support therapy for those who needs invasive or non-invasive oxygen therapy will be documented

CONTACTS AND LOCATIONS:
Locations (1):
- Nasr City Insurance Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No